CLINICAL TRIAL: NCT03782623
Title: Effect of Packed Red Blood Cell Transfusion on Eicosanoid Profiles in Plasma of Intensive Care Patients - a Pilot Study
Brief Title: Effect of Packed Red Blood Cell Transfusion on Eicosanoid Profiles in Plasma of Intensive Care Patients
Acronym: EICOTRANS-p
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment secondary to limited capacity during Covid-19 pandemic
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, PhD, Principle Investigator, Medical University of Vienna
Other Study IDs: 1595/2018
Record Dates: First submitted 2018-09-16; First posted 2018-12-20 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Anemia; Critical Illness; Lung Transplantation; Open Aortic Surgery
MeSH Terms: conditions — Anemia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intensive care patients after elective open aortic surgery
  Interventions: Diagnostic Test: Analysis of eicosanoid profile prior to and after PRBC transfusion
- Intensive care patients after bilateral lung transplantation
  Interventions: Diagnostic Test: Analysis of eicosanoid profile prior to and after PRBC transfusion
- Anesthetic intensive care patients, unplanned admission
  Interventions: Diagnostic Test: Analysis of eicosanoid profile prior to and after PRBC transfusion

INTERVENTIONS:
Diagnostic Test: Analysis of eicosanoid profile prior to and after PRBC transfusion — Using liquid chromatography-mass spectrometry to analyze the eicosanoid profile in patient plasma and aliquoted of the PRBCs prior to and after PRBC transfusion.

SUMMARY:
The main goal of this pilot study is to assess the time course of eicosanoid profiles in intensive care unit (ICU) patients requiring packed red blood cell (PRBC) transfusion. Moreover we will analyze the change of levels of eicosanoids in patient plasma prior and after a PRBC transfusion as well as its correlation with levels of eicosanoids in the transfused PRBCs. These data will then be used to determine the estimated effect size necessary for the planning of future larger studies. We hypothesize that transfusion of PRBCs will modulate the eicosanoid profile in ICU patients.

According to the Protocol filed with the Institutional Review Board of the Medical University of Vienna and patient's informed consent, subsequent sub analyses using samples of this study (e.g., determination of extracellular vesicles in PRBC samples and patient's plasma) will be performed.

ELIGIBILITY:
Exclusion Criteria:

* Age <18 years or >99 years
* Pregnancy
* <12h since last PRBC transfusion
* intake/administration of acetylsalicylic acid in groups 2 and 3
* intake/administration of cysteinyl leukotriene receptor antagonists (e.g. montelukast)
* intake/administration of celecoxib, etoricoxib, parecoxib, ibuprofen, diclofenac, and naproxen in all groups
* glucocorticoids given within 24h of transfusion in groups 1 and 3
* treatment with calcineurin inhibitors (e.g. tacrolimus) in groups 1 and 3
* treatment with alemtuzumab in groups 1 and 3
* administration of protamine for heparin reversal in groups 2 and 3

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: routine postoperative ICU patients after open aortic surgery Group 2: routine postoperative ICU patients with immunosuppression after lung transplantation Group 3: mixed postoperative ICU patients
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of plasma eicosanoid concentrations in ICU patients subjected to PRBC Transfusion at any time Point compared to baseline | 60 minutes prior to 90 minutes after packed red blood cell transfusion

SECONDARY OUTCOMES:
Changes of plasma eicosanoid profiles after PRBC transfusion compared to prior to PRBC transfusion in ICU patients | 60 minutes prior to 90 minutes after packed red blood cell transfusion
Correlation of plasma eicosanoid profiles in the transfused PRBCs and the change of their plasma levels in ICU patients | 60 minutes prior to 90 minutes after packed red blood cell transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raeven P, Karlhofer K, Sztulman LS, Brugger J, Hoetzenecker K, Domenig C, Leitner G, Posch M, Baron DM, Spittler A. Red blood cell transfusion-related dynamics of extracellular vesicles in intensive care patients: a prospective subanalysis. Sci Rep. 2024 Jan 9;14(1):911. doi: 10.1038/s41598-023-48251-w. PMID 38195728